CLINICAL TRIAL: NCT04565860
Title: Erciyes University Clinical Research Ethics Committee
Brief Title: Clinical Evaluation of Bulk-fill Composite Resins in Class II Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Nazire Nurdan Çakır, Assist. Prof Nurdan Çakır, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2015/281
Record Dates: First submitted 2020-09-15; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Dental Composite
Keywords: Bulk-fill composite; Incremental technique; Composite resin; FDI; USBHS

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- X-tra fil (bulk-filling) (X-traB) (Active Comparator): X-tra fil composite placed as bulk-filling
  Interventions: Other: Bulk-fill composite resin. (Dental Composite Resin Materials) (Dental filling materials)
- X-tra fil (incremental) (X-traI) (Active Comparator): X-tra fil composite placed as incremental
  Interventions: Other: Bulk-fill composite resin. (Dental Composite Resin Materials) (Dental filling materials)
- Filtek Bulk (bulk-filling) (FBB) (Active Comparator): Filtek Bulk composite placed as bulk-filling
  Interventions: Other: Bulk-fill composite resin. (Dental Composite Resin Materials) (Dental filling materials)
- Filtek Bulk (incremental) (FBI) (Active Comparator): Filtek Bulk composite placed as incremental
  Interventions: Other: Bulk-fill composite resin. (Dental Composite Resin Materials) (Dental filling materials)

INTERVENTIONS:
Other: Bulk-fill composite resin. (Dental Composite Resin Materials) (Dental filling materials) — Bulk-fill composites that were introduced in recent years are dental filling materials. Traditionally, the composite resins are placed in increments of 2 mm that are cured separately (incremental technique). Bulk-fill composites can be described as composites that are sufficiently polymerizable in a single layer up to 4 mm thick.
  In this study, each bulk-fill composite resin was used both in bulk-filing and incremental techniques for the same patient. The study set to 4 groups and 20 restorations in each group (a total of 80 restorations).
  Other Names: X-tra fil (Voco) bulk-fill composite resin. Filtek Bulk (3M ESPE) bulk-fill composite resin

SUMMARY:
Composite resins have been widely used in the last years to restore teeth due to increases in patients' esthetic expectations. Therefore optical and mechanical properties of composite resins were being developed day by day. Although there have been many in vitro studies about bulk-fill composite in the literature, the number of clinical trials is insufficient. Therefore, the aim of this study was to evaluate the clinical performance of bulk-fill composite about placement technique (bulk-filling and incremental techniques) in Class II carious lesions using the criteria of the World Dental Federation (FDI) and the United States Public Health Service (USPHS).

DETAILED DESCRIPTION:
Composite resins have been widely used in the last years to restore teeth due to increases in patients' esthetic expectations. Therefore optical and mechanical properties of composite resins were being developed day by day. Composite resin restorations have the main advantages such as conservative cavity preparation, preserving healthy dental tissue, and strengthening the remaining tooth structure. Furthermore, according to clinical studies, high clinical performance and good longevity have been reported. Traditionally, the composite resins are placed in increments of 2 mm that are cured separately (incremental technique. The incremental technique provides sufficient light penetration and monomer conversion. However, there are many disadvantages to the incremental technique. For instance, bonding failure, blood, or saliva contamination of between layers, the difficulty of application in limited access in small cavities, and to be time-consuming. Because of these, manufacturers have presented a "bulk-fill composites", which could be polymerized in a single layer up to 4-5 mm thick to the market. Bulk-fill composites can be described as composites that are sufficiently polymerizable in a single layer up to 4 mm thick. Bulk-fill composites that were introduced in recent years can be manipulated faster and more convenient in the cavity compared to conventional hybrid composites. In addition, these materials present good mechanical properties such as marginal adaptation, sealing properties, fracture strength, wear-resistance, and long-term clinical success. Clinical studies are required to clearly describe the clinical behavior of the materials. Although there have been many in vitro studies about bulk-fill composite in the literature, the number of clinical trials is insufficient. Therefore, the aim of this study was to evaluate the clinical performance of bulk-fill composite about placement technique (bulk-filling and incremental techniques) in Class II carious lesions using the criteria of the World Dental Federation (FDI) and the United States Public Health Service (USPHS)

ELIGIBILITY:
Inclusion Criteria:

* At least 4 Class-II caries lesions
* Good health
* Acceptable level of oral hygiene

Exclusion Criteria:

* Did not have four caries lesions at least
* Did not have Class-II caries lesions
* Deep caries reaching the pulp
* The patients are not 18-20 years old
* Bruxism
* Periodontal disease
* Refused to participate

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical performance of bulk-fill composite about placement technique (bulk-filling and incremental) in Class II carious lesions using FDI and USPHS criteria. | Two-year
  FDI; The World Dental Federation. USPHS; The United States Public Health Service. The 2-year results of the restorations were evaluated with the FDI and USPHS criteria. Two calibrated observers who were blinded to the objective of this study performed the evaluations.
Evaluation of the clinical performance of bulk-fill composite about placement technique (bulk-filling and incremental) in Class II carious lesions using FDI and USPHS criteria. | Four-year
  FDI; The World Dental Federation. USPHS; The United States Public Health Service. The 4-year results of the restorations were evaluated with the FDI and USPHS criteria. Two calibrated observers who were blinded to the objective of this study performed the evaluations.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided